CLINICAL TRIAL: NCT06232980
Title: Evaluation of Observer Alertness/Sedation Score (OAA/S) and Bispectral Index (BIS) Parameters for Induction of General Anesthesia With Propofol in Geriatric Patients
Brief Title: The Use of Sedation Score and Bispectral Index for Induction in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UfukTakak1
Record Dates: First submitted 2024-01-10; First posted 2024-01-31 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: E03.155.253; Bispectral Index Monitor; Hypotension
Keywords: geriatric anesthesia; bispectral index monitor; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Group O: HR, SAB, DAB, OAB, SpO2, and BIS values will be recorded at 2-minute intervals for 14 minutes. A standard initial dose of 1.5 mg/kg of propofol and an infusion rate of 100 mg/min will be applied. An additional 20 mg of propofol will be administered every 30 seconds until the Observer's Assessment of Alertness/Sedation (OAA/S) score reaches 1.
  Group B: HR, SAB, DAB, OAB, SpO2, and BIS values will be recorded at 2-minute intervals for 14 minutes. The BIS index will be evaluated every 30 seconds. The initial dose and infusion rate will be applied as in Group O, with the target index in the BIS group being 40-60. An additional dose of 20 mg will be planned every 30 seconds until the target index is reached.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthesia induction group guided by BIS in geriatric patients. (Active Comparator): The BIS index will be evaluated every 30 seconds. The initial dose and infusion rate will be applied as 1.5 mg/kg and 100 mg/min, respectively. In the BIS group, the target index is set between 40-60, and additional doses of 20 mg will be planned every 30 seconds until reaching this target index.
  Interventions: Procedure: urological surgical intervention
- Observer's Alertness/Sedation Score-guided induction group in geriatric patients. (Active Comparator): The initial dose will be applied as 1.5 mg/kg, and the infusion rate will be 100 mg/min. An additional 20 mg of propofol will be administered every 30 seconds until the Observer's Assessment of Alertness/Sedation (OAA/S) score reaches 1.
  Interventions: Procedure: urological surgical intervention

INTERVENTIONS:
Procedure: urological surgical intervention — Anesthesia induction will be performed with propofol, and ventilation will be maintained with a laryngeal mask for urological surgical procedures.

SUMMARY:
The main objective of this clinical study is to determine the effectiveness of BIS-guided propofol administration in avoiding hypotension during propofol induction in geriatric patients. The primary question it aims to answer is whether the mean arterial pressure can be maintained above 60mmHg with BIS-guided propofol induction. For this purpose, the observer's alertness sedation score will be compared with bispectral index-guided inductions.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the effectiveness of BIS-guided propofol administration to avoid hypotension in propofol induction in geriatric patients. Mean arterial pressure (MAP) below 60 mmHg is defined as hypotension. The secondary aims include finding the differences between the entry MAP and the MAP at each measurement, determining the difference between the entry MAP and the lowest MAP, determining the ratio of hypotensive and normotensive MAP measurements, determining the number of patients with severe hypotension (MAP<50 mmHg), determining the number of patients receiving vasopressor therapy and drug dosage, determining the number of patients who underwent Trendelenburg, and those who developed tachycardia (HR>100/min), determining the number of patients who developed hypertension (MAP>140), and finding the correlation between BIS values and MAP. T.R. In the Ministry of Health Ankara City Hospital Urology Operating Room, general anesthesia will be applied, and ventilation will be provided with LMA as two different approaches for patients over 65 years of age; By evaluating OAA/S-based propofol induction and BIS-guided propofol inductions, the investigators aim to investigate whether the use of BIS reduces the risk of developing hypotension by reducing the propofol dose in anesthesia induction. T.R. After receiving ethics committee approval at the Ministry of Health Ankara City Hospital Urology Operating Room, 122 patients over the age of 65 who will receive general anesthesia and ventilation with a laryngeal mask (LMA) under elective conditions will be included in the study.

The study will be designed as a prospective randomized controlled trial. A total of 122 patients undergoing elective surgery in the urology operating room will be divided into two groups, Group O and Group B, using computer-assisted randomization. Group O will undergo an anesthesia induction guided by OAA/S, while Group B will undergo a general anesthesia induction guided by BIS.

After being admitted to the operating room, Group O will have recorded heart rate (HR) in beats per minute, systolic arterial blood pressure (SAB) in mmHg, diastolic arterial blood pressure (DAB) in mmHg, mean arterial blood pressure (OAB) in mmHg, peripheral oxygen saturation (SpO2), and BIS values. Four milliliters per kilogram of appropriate balanced crystalloid solution will be administered 2 minutes after the start, and HR, SAB, DAB, OAB, SpO2, and BIS values will be reevaluated. These values will be recorded every 2 minutes for 14 minutes. Premedication will not be administered, and anesthesia induction will begin with 1 mcg/kg fentanyl. Many commonly used anesthesia induction agents, including propofol, can cause significant and even life-threatening drops in blood pressure, respiratory depression, and other adverse events. The dose ranges of propofol decrease with age, leading to the FDA's recommendation to reduce the induction dose from 2-2.5 mg/kg in geriatric patients to 1-1.5 mg/kg. In the clinic, a standard initial dose of 1.5 mg/kg of propofol and an infusion rate of 100 mg/min are applied in geriatric patients. The initial dose for both groups will be 1.5 mg/kg, and the infusion rate will be 100 mg/min. An additional 20 mg of propofol will be administered every 30 seconds until the Observer's Assessment of Alertness/Sedation (OAA/S) score is 1. In case of hypotension, the management of hypotension (vasopressor treatment, Trendelenburg position, fluid loading) is left to the discretion of the responsible anesthesiologist. Anesthesia maintenance will be provided with volatile anesthetics. At the end of the procedure, hemodynamic parameters (SAB, DAB, OAB, HR, SpO2), BIS values, Observer's Assessment of Alertness/Sedation Scale (OASS), time to reach OAA/S 1, anesthesia induction drug and doses, hypotension treatment, and airway equipment placement time will be recorded.

Upon admission to the operating room, Group B will have recorded heart rate (HR) in beats per minute, systolic arterial blood pressure (SAB) in mmHg, diastolic arterial blood pressure (DAB) in mmHg, mean arterial blood pressure (OAB) in mmHg, peripheral oxygen saturation (SpO2), and BIS values. Four milliliters per kilogram of appropriate balanced crystalloid solution will be administered 2 minutes after the start, and HR, SAB, DAB, OAB, SpO2, and BIS values will be reevaluated. These values will be recorded every 2 minutes for 14 minutes. Premedication will not be administered, and anesthesia induction will begin with 1 mcg/kg fentanyl. The time delay between propofol injection and the decrease in BIS index depends on the drug transition time (from the injection site to the effect site) and the index calculation time. Time delays between 14 and 155 seconds have been reported for the BIS index. In the study, the BIS index will be evaluated every 30 seconds. The initial dose and infusion rate will be applied as in Group O, with the target index in the BIS group being 40-60. An additional dose of 20 mg will be planned every 30 seconds until the target index is reached. In case of hypotension, the management of hypotension (vasopressor treatment, Trendelenburg position, fluid loading) is left to the discretion of the responsible anesthesiologist. At the end of the procedure, hemodynamic parameters (SAB, DAB, OAB, HR, SpO2), BIS values, time to reach BIS <60, Observer's Assessment of Alertness/Sedation Scale (OASS), anesthesia induction drug and doses, hypotension treatment, and airway equipment placement time will be recorded.

The sample size calculation was performed using MedCalc 15.8 (MedCalc Software bvba, Ostend, Belgium). It was determined that a minimum of 122 patients (61 + 61) is sufficient for P1 = 0.6, P2 = 0.3, α = 0.05, and a power of 90% (1-β).

ELIGIBILITY:
Inclusion Criteria:

* T.R. Patients aged 65 and over who will undergo elective surgery under general anesthesia in the Urology Operating Room of the Ministry of Health Ankara City Hospital

Exclusion Criteria:

* Being under 65 years old
* Those who do not have the ability to read, understand and sign the consent form
* Hemodynamically unstable patients
* Those who have contraindications to anesthetic drugs
* Patients who do not want to participate in the study
* Patients with advanced dementia
* Emergency surgical procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Use of BIS for preventing hypotension (mean arterial pressure (MAP) <60 mmHg) during propofol induction in geriatric patients | The mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes.

SECONDARY OUTCOMES:
Find the differences between the input MAP and the MAP at each measurement | The mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes, and the differences between the entry MAP and the MAP at each measurement will be determined.
Find the difference between input MAP and lowest MAP | Mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes, and the difference between the entry MAP and the lowest MAP will be determined.
To determine the ratio of hypotensive and normotensive MAP measurements | The mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes, and the ratio of hypotensive to normotensive MAP measurements will be determined.
To determine the number of patients with severe hypotension (MAP<50 mmHg) | Mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes, and the number of patients experiencing severe hypotension (MAP<50 mmHg) will be determined.
To determine the number of patients receiving vasopressor therapy and the drug dosage | The mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes, and the number of patients developing hypotension receiving vasopressor therapy, along with the drug dosage, will be determined.
To determine the number of patients who underwent Trendelenburg | The mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes, and the number of patients with hypotension who undergo Trendelenburg positioning will be determined.
To determine the number of patients who developed tachycardia (HR>100/min) | Heart rate will be recorded at 2-minute intervals for a duration of 14 minutes, and the number of patients developing tachycardia (heart rate >100 beats per minute) during this period will be determined.
To determine the number of patients who developed hypertension (MAP>140) | The mean arterial pressure (MAP) will be recorded at 2-minute intervals for a duration of 14 minutes, and the number of patients developing hypertension (MAP >140 mmHg) will be determined.
Finding the correlation between BIS values and MAP | MAP, bispectral index, and the duration until the bispectral index reaches the range of 40-60 will be recorded at 2-minute intervals for a duration of 14 minutes. The correlation between bispectral index and MAP.

CONTACTS AND LOCATIONS:
Overall Officials: ayşe lafçı, Principal Investigator — ankara bilkent city hospital, anesthesiology and reanimation clinic
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Devinney MJ, Berger M. Goldilocks and propofol dosage in older adults: Too much, too little, or just right? J Am Geriatr Soc. 2021 Aug;69(8):2106-2109. doi: 10.1111/jgs.17221. Epub 2021 May 8. No abstract available. PMID 33964173
- [Result] Rusch D, Arndt C, Eberhart L, Tappert S, Nageldick D, Wulf H. Bispectral index to guide induction of anesthesia: a randomized controlled study. BMC Anesthesiol. 2018 Jun 15;18(1):66. doi: 10.1186/s12871-018-0522-8. PMID 29902969
- [Result] Pilge S, Zanner R, Schneider G, Blum J, Kreuzer M, Kochs EF. Time delay of index calculation: analysis of cerebral state, bispectral, and narcotrend indices. Anesthesiology. 2006 Mar;104(3):488-94. doi: 10.1097/00000542-200603000-00016. PMID 16508396
- [Result] Gurses E, Sungurtekin H, Tomatir E, Dogan H. Assessing propofol induction of anesthesia dose using bispectral index analysis. Anesth Analg. 2004 Jan;98(1):128-131. doi: 10.1213/01.ANE.0000090314.43496.1D. PMID 14693603
- [Result] Schmidt GN, Bischoff P, Standl T, Lankenau G, Hilbert M, Schulte Am Esch J. Comparative evaluation of Narcotrend, Bispectral Index, and classical electroencephalographic variables during induction, maintenance, and emergence of a propofol/remifentanil anesthesia. Anesth Analg. 2004 May;98(5):1346-53, table of contents. doi: 10.1213/01.ane.0000111209.44119.30. PMID 15105213
- [Result] Chen L, Lu K, Luo T, Liang H, Gui Y, Jin S. Observer's Assessment of Alertness/Sedation-based titration reduces propofol consumption and incidence of hypotension during general anesthesia induction: A randomized controlled trial. Sci Prog. 2021 Oct;104(4):368504211052354. doi: 10.1177/00368504211052354. PMID 34825617